CLINICAL TRIAL: NCT03394339
Title: Relation of Fruit and Vegetable Sources With Cardiovascular Outcomes: A Systematic Review and Meta-analysis of Prospective Cohort Studies.
Brief Title: Meta-analysis of Fruit and Vegetable Sources and Cardiovascular Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: CIHR-FRU VEG & CVD 2017
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: CHD - Coronary Heart Disease; CVD - Cerebrovascular Disease; Stroke
Keywords: Systematic review and meta-anaylsis; Evidence-based nutrition (EBN); Dietary guidelines; Fruit; Vegetables
MeSH Terms: conditions — Coronary Artery Disease; Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fruit and vegetables are a cornerstone of healthy dietary patterns and dietary guidelines worldwide. The supporting evidence, however, is largely derived from observational studies of protective associations with cardiovascular disease (CVD) in health-conscious populations or from randomized trials of the effect of specific fruit or vegetable derived nutrients on CVD risk factors. A growing body of literature has influenced a shift away from a focus on single nutrients to a focus on whole foods and dietary patterns. To what extent fruit and vegetables should contribute to dietary patterns for cardiovascular health and whether specific types of fruit or vegetables should be recommended is unclear. Although previous systematic reviews and meta-analyses have elucidated the association between the intake of total and some specific fruit and vegetables with cardiovascular outcomes, a comprehensive synthesis comparing the certainty of the evidence for the different types of fruit and vegetables in relation to a range of cardiovascular outcomes has yet to be completed. We propose to conduct a systematic review and meta-analysis of the available prospective cohort studies using the Grading of Recommendations Assessment, Development, and Evaluation (GRADE) approach to assess the association between different types of fruit and vegetables and different cardiovascular outcomes that include CVD, coronary heart disease [CHD], and stroke incidence and mortality.

DETAILED DESCRIPTION:
Background:

A high intake of fruit and vegetables is a common trait among healthy dietary patterns and a cornerstone of nutrition interventions for cardiovascular disease (CVD) prevention. There is an international consensus that at least 5 servings per day of fruit and vegetables is beneficial to overall population health (WHO, 2003). This guidance, however, is largely founded on observational studies showing protective associations of high intakes of fruit and vegetables with CVD in health-conscious individuals (Reddy and Katan, 2004). Recommendations to consume specific types of fruit and vegetables, such as citrus fruit and green leafy vegetables, have been established mainly on the association of isolated nutrients with CVD risk reduction in observational studies or the effect of isolated nutrients on CVD risk factors in small randomized trials (Katamay et al., 2007). Given its prominence in dietary guidelines, there is a need to determine the extent of CVD risk reduction that may be attributed to the consumption of fruit and vegetables. As guidelines are shifting away from a focus on single nutrients to a focus on whole foods and dietary patterns and achieving adequate intakes continue to be a challenge worldwide and (Hall et al., 2009), there is also an advantage in establishing which types of fruit and vegetables are associated with the greatest protection in CVD incidence and mortality per serving. Although several systematic reviews and meta-analyses of prospective cohort studies have demonstrated protective associations between the intake of total fruit and vegetables and CVD risk (Aune et al., 2017; Zhan et al., 2017; Gan et al., 2015; Wang et al, 2014; Hu et al., 2007; He et al., 2007; Dauchet et al., 2006), few have focused on specific fruit and vegetables or explored a range of cardiovascular outcomes which may have different etiologies. Several large prospective cohort studies have recently been published which may strengthen the certainty of the evidence by increasing the number of observations for the relationship between different fruit and vegetables exposures and different cardiovascular outcomes. We propose to build and expand on the exiting systematic reviews and meta-analyses by conducting a comprehensive synthesis of prospective cohort studies comparing the certainty of the evidence for the different types of fruit and vegetables in relation to a range of cardiovascular outcomes.

Objective:

To conduct a systematic review and meta-analysis of the available prospective cohort studies using the Grading of Recommendations Assessment, Development, and Evaluation (GRADE) approach to assess the association between different types of fruit and vegetables and different cardiovascular outcomes including CVD, CHD, and stroke incidence and mortality.

Design:

The conduct of the proposed systematic review and meta-analysis will follow the Cochrane handbook for systematic reviews of interventions and the GRADE handbook for grading the certainty of the evidence and the strength of recommendations using the GRADE approach. The reporting will follow the Meta-Analysis Of Observational Studies in Epidemiology (MOOSE) and the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA) statements.

Data Sources:

MEDLINE, Embase, and the Cochrane Central Register of Controlled Trials (CENTRAL) will be searched using relevant search terms. Search of databases will be supplemented by manual searches of bibliographies.

Study Selection:

Prospective cohort studies exploring the relation of fruit and/or vegetable intake to incident cardiovascular disease for a minimum follow-up time of 1 year will be included.

Data extraction:

Two independent reviewers will extract relevant information including study design, sample size, subject characteristics, exposure form (i.e. total fruit and vegetables, citrus fruit, green leafy vegetables, etc.), duration/person-years of follow-up, adjustments of models and risk ratios for clinical outcomes derived from clinical event data across quantiles of exposure. Any disagreements will be reconciled by consensus with arbitration by the Principal Investigator.

Risk of bias:

Risk of bias (ROB) will be assessed by two independent reviewers using the Newcastle-Ottawa Scale (NOS). Up to 9 points can be awarded based on cohort selection (max 4 points), the comparability of cohort design and analysis (max 4 points), and adequacy of the outcome measures (max 3 points). Studies that receive ≥6 points will be considered as higher quality. Again, any disagreements will be reconciled by consensus with arbitration by the Principal Investigator.

Outcomes:

We will assess 6 outcomes: CVD incidence and mortality, CHD incidence and mortality, and stroke incidence and mortality.

Data Synthesis:

We will pool the natural log-transformed relative risks for the 6 cardiovascular outcomes using the inverse variance method with random effects models with data expressed as risk ratios (RR) with 95% confidence intervals (CIs). Analyses will be conducted by extreme quantiles analyses, comparing the highest with the lowest (reference) level of exposure. Data will also be scaled to allow for per serving/day analyses. Between-study heterogeneity will be assessed by the Cochran Q test and quantified by the I2 statistic with significance at P<0.1. An I2≥50% and P<0.1 will be considered as evidence of substantial heterogeneity. Sensitivity analyses and a priori subgroup analyses will be undertaken to explore sources of heterogeneity. Sensitivity analyses will include the systematic removal of included cohorts with the recalculation of summary estimates. A priori subgroup analyses will be conducted when ≥10 cohort comparisons are available by age, sex, location of cohort, follow-up duration, dietary assessment tool, risk of bias (NOS score). A separate subgroup analysis will also be conducted by each domain of risk of bias by NOS. Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. Dose-response analyses will be undertaken using random-effects generalized least squares trend estimation models (GLST) to assess linear relationships and spline curve modeling (the MKSPLINE procedure) to assess non-linear relationships. If ≥10 cohort comparisons are available, then publication bias will be assessed by visual inspection of funnel plots and formal testing with the Egger and Begg tests at a significance level of p≤ 0.10. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Grading the Evidence:

The Grading of Recommendations Assessment, Development and Evaluation (GRADE) method will be used to assess the overall certainty of the evidence for each of the cardiovascular outcomes. This system grades the evidence as "high quality", "moderate quality", "low quality", or "very low quality". Observational studies including prospective cohort studies start at a "low quality" and then can be downgraded or upgraded based on established criteria. Criteria to downgrade will include study limitations (weight of studies show risk of bias by NOS), inconsistency (substantial unexplained inter-study heterogeneity, I2>50%, P<0.10), indirectness (presence of factors relating to the population, exposures, and outcomes that limit generalizability), imprecision (95% CI are wide or cross a minimally important difference of 5% [RR 0.95- 1.05]), and publication bias (significant evidence of publication bias or small-study effects). Criteria to upgrade will include a large magnitude effect (RR>2 or RR<0.5 in the absence of plausible confounders), a dose-response gradient, and attenuation by plausible confounding effects.

Knowledge translation plan:

The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, physical activity, lifestyle modification, obesity, diabetes, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined.

Significance:

The study will aid in establishing a stronger evidence-base to determine the extent to which a high fruit and vegetable intake may be associated with reduction in incident CVD. It may also bring to light categories of fruits and/or vegetables that could provide additional benefit in CVD prevention.

References:

World Health Organization. (2003). Fruit and Vegetable Promotion Initiative - report of the meeting. Geneva.

Reddy KS and Katan MB. (2004). Diet, nutrition and the prevention of hypertension and cardiovascular disease. Public Health Nutrition. 7(1A): 167-186

Katamay SW, Esslinger KA, Vigneault M, et al. (2007) Nutrition Reviews. 65(4): 155-166.

Hall JN, Moore S, Harper SB, et al. (2009). Global variability in fruit and vegetable consumption. American Journal of Preventative Medicine. 36:402-409

Aune D, Giovannucci E, Boffetta P, et al. (2017). Fruit and vegetable intake and the risk of cardiovascular disease, total cancer and all-cause mortality - a systematic review and dose-response meta-analysis of prospective studies. International Journal of Epidemiology. 1-28

Zhan J, Liu Y, Cai L, et al. (2017). Fruit and vegetable consumption and risk of cardiovascular disease: A meta-anaylsis of prospective cohort studies. Critical Reviews in Food Science and Nutrition. 57(8):1650-1663

Gan Y, Tong X, Liqing L, et al. (2015). Consumption of fruit and vegetable and risk of coronary heart disease: A meta-analysis of prospective cohort studies. International Journal of Cardiology. 183: 129-137

Wang X, Ouyang Y, Liu J, et al. (2014). Fruit and vegetable consumption and mortality from all causes, cardiovascular disease, and cancer: systematic review and dose-response meta-analysis of prospective cohort studies. British Medical Journal. 349

Hu D, Hunag J, Wang Y, et al. (2014). Fruits and vegetables consumption and risk of stroke: A meta-analysis of prospective cohort studies. Stroke. 45: 1613-1619

He FG, Nowson CA, Lucas M et al. (2007). Increased consumption of fruit and vegetables is related to reduced risk of coronary heart disease: meta-analysis of cohort studies. Journal of Human Hypertension. 21:717-728

He FJ, Nowson CA and MacGregor GA. (2006). Fruit and vegetable consumption and stroke: a meta-analysis of cohort studies. Lancet: 367:320-326.

Dauchet L, Amouyel P, Hereberg S, et al. (2006). Fruit and vegetable consumption and risk of coronary heart disease: A meta-analyses of cohort studies. The Journal of Nutrition. 136: 2588-2593.

ELIGIBILITY:
Inclusion Criteria:

* Prospective cohort studies or case-cohort studies
* Duration >= 1 year
* Assessment of the exposure of fruit and/or vegetables
* Ascertainment of viable data by level of exposure

Exclusion Criteria:

* Ecological, cross-sectional, and retrospective observational studies, clinical trials, and non-human studies
* Duration < 1 year
* No assessment of exposures of fruit or vegetables
* No ascertainment viable clinical outcome data by level of exposure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Varied
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease (CVD) | 1 year follow-up
  Risk ratios for CVD incidence and mortality
Coronary heat disease (CHD) | 1 year follow-up
  Risk ratios for CHD incidence and mortality
Stroke | 1 year follow-up
  Rsk ratios for stroke incidence and mortality

CONTACTS AND LOCATIONS:
Overall Officials: John Sievenpiper, MD, PhD, FRCPC, Principal Investigator — Department of Nutritional Sciences, Faculty of Medicine, University of Toronto and Clinical Nutrition and Risk Factor Modification Centre and Toronto 3D Knowledge Institute and Clinical Trials Unit, St. Michael's Hospital; Sonia Blanco Mejia, MD, Study Director — Clinical Nutrition and Risk Factor Modifcation Centre and Toronto 3D Knowledge Institute and Clinical Trials Unit, St. Michael's Hosptial
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All data will be available in the publication

REFERENCES:
- [Derived] Zurbau A, Au-Yeung F, Blanco Mejia S, Khan TA, Vuksan V, Jovanovski E, Leiter LA, Kendall CWC, Jenkins DJA, Sievenpiper JL. Relation of Different Fruit and Vegetable Sources With Incident Cardiovascular Outcomes: A Systematic Review and Meta-Analysis of Prospective Cohort Studies. J Am Heart Assoc. 2020 Oct 20;9(19):e017728. doi: 10.1161/JAHA.120.017728. Epub 2020 Oct 1. PMID 33000670